CLINICAL TRIAL: NCT06746662
Title: The Effect of Hypnobreastfeeding Philosophy-Based Counseling on Breastfeeding Self-Efficacy and Breastfeeding Success in Adolescent Pregnant Women
Brief Title: The Effect of Hypno-Lactation Counseling on Breastfeeding Self-Efficacy and Breastfeeding Success in Adolescent Pregnant Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, İpek TURAN, Student, Cukurova University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: ipekt1
Record Dates: First submitted 2024-12-03; First posted 2024-12-24 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Pregnant Women
Keywords: Hypnobreastfeeding; breastfeeding self-efficacy; breast-feeding; Adolescent pregnant; breastfeeding success
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Hypno-breastfeeding Education Group
  A counseling program based on hypno-breastfeeding philosophy, where 4-week education content will be presented to pregnant adolescents in their 28-30th week of pregnancy and applications will be made, will be implemented with 4 sessions and 6 follow-ups. A breastfeeding education booklet (Appendix 6) will be prepared in the implementation of the counseling service. Each session will last an average of 1 hour. The training sessions will be conducted face-to-face. The average number of pregnant women in each follow-up will consist of 3-5 people. During and after the training processes, pregnant women will be provided with regular information based on hypno-breastfeeding philosophy, affirmation, relaxation techniques and meditation materials (Appendix 6) and counseling based on hypno-breastfeeding philosophy.
  First follow-up (28-30th week of pregnancy - first encounter): This midwifery intervention will be performed on pregnant women in a suitable roo
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counseling based on the philosophy of hypnobreastfeeding (Experimental): Hypno-breastfeeding is a method that involves a natural effort to use subconscious energy so that the breastfeeding process can proceed comfortably and smoothly and the mother can produce enough breast milk for the baby's growth and development needs (AIMI, 2010; Sofiyanti et al., 2019). With hypno-breastfeeding, the breastfeeding process takes place comfortably and the mother subconsciously registers that breastfeeding is a natural and comfortable process (Sembırıng, 2017; Altıparmak, 2021; Kilçi Erciyas and Sevil, 2021). In the philosophy of hypno-breastfeeding, positive schemas for breastfeeding are created in the subconscious. By focusing on the use of the primitive brain, the stimulation of the neocortex with unnecessary information and stimuli is avoided (Aluş Tokat and Gökçe İsbir, 2023). This technique, which helps to facilitate a holistic look at the mind, body and soul of breastfeeding mothers, allows the mother to be more relaxed, calm and comfortable during breastfeeding
  Interventions: Behavioral: Hypnobreastfeeding training and consultancy
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Hypnobreastfeeding training and consultancy — Hypno-breastfeeding Education Group
  A counseling program based on hypno-breastfeeding philosophy, where 4-week education content will be presented to pregnant adolescents in their 28-30th week of pregnancy and applications will be made, will be implemented with 4 sessions and 6 follow-up
  Arms: Counseling based on the philosophy of hypnobreastfeeding

SUMMARY:
This study aimed to investigate the effects of counseling based on hypno-breastfeeding philosophy on breastfeeding self-efficacy and breastfeeding success in pregnant adolescents.

Research Hypotheses H1a: The intervention group's breastfeeding self-efficacy after hypno-breastfeeding counseling is different from the control group.

H1b: The intervention group's breastfeeding success after hypno-breastfeeding counseling is different from the control group.

This thesis is a randomized controlled experimental study. The study is planned to be conducted with two parallel groups, namely the intervention and control groups. Hypno-breastfeeding training will be applied to the intervention group, and standard breastfeeding training will be applied to the control group. The study will be conducted with pregnant adolescents who applied to the pregnancy clinic of Adıyaman University Training and Research Hospital between December 2024 and April 2025.

DETAILED DESCRIPTION:
This study aimed to investigate the effects of counseling based on hypno-breastfeeding philosophy on breastfeeding self-efficacy and breastfeeding success in pregnant adolescents.

Place, type and time of the study This thesis study is a randomized controlled experimental study. The study is planned to be conducted with two parallel groups, the intervention and control groups. Hypno-breastfeeding training will be applied to the intervention group, and standard breastfeeding training will be applied to the control group. The study will be conducted with pregnant adolescents who applied to the pregnancy clinic of Adıyaman University Education and Research Hospital between December 2024 and April 2025.The Universe and Sample of the Study: The universe of the study consists of pregnant adolescents registered at the 400-bed Adıyaman University Training and Research Hospital.

Data Collection Tools Data will be collected using the Personal Information Form (Appendix 1), Breastfeeding Self-Efficacy Scale-Short Form (Appendix 2) and Breastfeeding Diagnostic Scale (LATCH) (Appendix 3) prepared by the researchers in line with the literature.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 16-19,
* Single pregnancy,
* Primiparous,
* Planning a normal vaginal birth,
* In the last trimester of pregnancy,
* No communication problems,
* Can speak and understand Turkish,
* Can read and write, as the scales must be filled out by the individual,
* No condition preventing breastfeeding,
* Not receiving any training/counseling regarding breastfeeding during pregnancy

Exclusion Criteria:

* Women who have been diagnosed with a psychiatric disorder,
* Complications in the mother and baby (chronic disease in the mother that prevents breastfeeding; diabetes, hypertension, etc. fetal anomalies in the fetus, postpartum discomfort that will prevent breastfeeding),
* Women who develop a health problem during pregnancy during the training process,
* Women who want to withdraw from the study voluntarily
* Women who have any disability (hearing impairment, etc.) will be excluded from the study.

Ages: 16 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Adolescent pregnant women
Enrollment: 60 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy | Baseline, 4 week, and after the labour
  The first form of the scale developed by Dennis and Faux was designed with 33 items, but after a second study, Dennis revised the scale and created a short form of 14 items (5). The Turkish validity and reliability study of the scale was conducted by Aluş Tokat and colleagues (6). The scale can be applied in the prenatal and postnatal periods and measures how adequate women feel about breastfeeding. The items of the five-point Likert-type scale are scored as not at all sure (1), not very sure (2), sometimes sure (3), sure (4), very sure (5). The lowest score that can be obtained from the entire evaluation scores of the scale is 14 and the highest score is 70. A low total score obtained from the scale indicates that the perception of breastfeeding self-efficacy is low.

SECONDARY OUTCOMES:
Breastfeeding Success | Baseline, 4 week, and after the labour
  The LATCH breastfeeding diagnosis and assessment scale is a diagnostic method used to assess breastfeeding success, first created in 1986 by resembling the APGAR scoring system in terms of scoring method . The average application time varies between 7-10 minutes. This measurement tool was developed to objectively diagnose breastfeeding, identify breastfeeding problems, create a common language among healthcare professionals and to be used in research (to determine breastfeeding success in longitudinal studies) . It consists of five evaluation criteria, and the abbreviation of the first letters of the English equivalents of these criteria constitutes the name of the scale.
  Each item is evaluated between 0-2 points. The highest total score that can be obtained is 10, and a high score means a high breastfeeding success.

IPD SHARING:
Plan to Share IPD: No